CLINICAL TRIAL: NCT04434677
Title: Comparative Study Between Hypofractionation And Ultra-Hypofractionation In Adjuvant Radiotherapy For Breast Cancer
Brief Title: Hypofractionation And Ultra-Hypofractionation In Adjuvant Radiotherapy For Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0201263
Record Dates: First submitted 2020-05-29; First posted 2020-06-17 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: radiotherapy; hypofractionation; ultrahypofractionation; 5 fractions
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionation (Active Comparator): Control arm:patients who will receive standard 40.05 Gray (2.67 Gy/ fx) over 15 fractions with or without boost over 3 weeks
  Interventions: Radiation: Hypofractionation
- Ultrahypofractionation (Experimental): Experimental arm: Patients who will receive 26 Gray (5.2 Gy/fx) over 5 fractions over 1.5 weeks
  Interventions: Radiation: ultraHypofractionation

INTERVENTIONS:
Radiation: Hypofractionation — 3D conformal Radiotherapy whole breast irradiation +- Supraclavicular fossa using Linear Machine (6-15 MV energy) 40.05 Gray (2.67 Gy/ fx) over 15 fractions with or without boost over 3 weeks
  Arms: Hypofractionation
Radiation: ultraHypofractionation — 3D conformal Radiotherapy whole breast irradiation +- Supraclavicular fossa using Linear Machine (6-15 MV energy) 26 Gray (5.2 Gy/fx) over 5 fractions over 1.5 weeks
  Arms: Ultrahypofractionation

SUMMARY:
Prospective randomized study comparing 5 fractions in alternative days to standard 15 fractions regarding effectiveness and feasibility during adjuvant treatment in breast caner patients aged above 50 years

DETAILED DESCRIPTION:
In Alexandria, the number of working linear machines are limited with overcrowded waiting list which lead to prolongation of overall treatment time and delay in starting radiotherapy. Providing the available data, Principle investigator is conducting this study in parallel with fast forward protocol to provide an alternative cost effective approach to patients.

The rationale behind hypofractionation depends mainly on the alpha beta ratio (α/β) and the overall treatment time. In Breast cancer the ratio is around 4 which is slightly lower than other tumors such as head and neck. The lower the ratio the higher the dose per fraction is needed to compensate slower proliferating tumors. Also, the overall treatment time could affect the local recurrence of breast cancer which is increased with long duration of treatment.

This study will include at least 100 patients with non metastatic histologically proved breast cancer who are indicated for adjuvant radiotherapy.

The patients will be randomized into two arms:

* Control arm: will include 50 patients who will receive standard 40.05 Gray (2.67 Gy/fx) over 15 fractions with or without boost over 3 weeks biologically effective dose (BED) for early and late effect equal 50.74.Gy10 and 75.69 Gy3 respectively.
* Experimental arm: will include 50 patients who will receive 26 Gray (5.2 Gy/fx) over 5 fractions over 1.5 weeks with BED for early and late effect equal 39.52 Gy10 and 71.07 Gy3 respectively

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50 years old.
* Informed consent.
* Either breast conservative surgery or mastectomy.
* Invasive breast cancer with p T1-3, p N0-2.
* Non metastatic breast cancer proven by clinical examinations and imaging (X-ray chest and ultrasound or CT scan chest and abdomen).

Exclusion Criteria:

* Evidence of distant metastases.
* Prior irradiation.
* Inflammatory breast cancer.
* Tumor with T4 (skin nodules or fixed to chest wall or ulceration).
* Tumor with positive margins.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-06-28 (Estimated); Study Completion 2021-06-28 (Estimated)

PRIMARY OUTCOMES:
Rate of Acute grade 2 or higher toxicity (NCI-CTCAE) | Start of treatment till 3 months from end of treatment
  Each patient will be assessed weekly during radiotherapy and monthly for three months post radiotherapy to assess acute toxicity and will be documented according to Common Terminology Criteria for adverse events (CTCAE)
Rate of chronic Toxicity grade 2 or higher (NCI-CTCAE) | Before start treatment and from 6 months after finishing treatment every 6 months up to average 2 years
  Each patient will be assessed before treatment and at 6 , 12 , 24 months for chronic toxicity Criteria for adverse events (CTCAE)
Rate of Ipsilateral local tumor recurrence | 1 to 2 years
  Local recurrence proved by image and biopsy
Compliance to treatment (number of interrupted days of radiation) | Start treatment till end of treatment (2 weeks in arm one and 3 weeks in arm2)
  Treatment interruptions of planned cycles

SECONDARY OUTCOMES:
Overall survival | From date of diagnosis up to average 2 years
  the percentage of people in a study or treatment group who are alive two years after the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf M El-Enbaby, Prof, Principal Investigator — Alexandria University
Locations (1):
- ACOD, Alexandria, Egypt